CLINICAL TRIAL: NCT01170078
Title: A Phase 1 Study Comparing the Pharmacokinetics of Epoetin Hospira and Epoetin Alfa (Amgen) When Administered Intravenously in Patients With Chronic Renal Failure Requiring Hemodialysis and Receiving Epoetin Maintenance Treatment
Brief Title: A Study Comparing the Effects of Epoetin Hospira and Epogen/Epoetin Alfa (Amgen) When Administered IV in Patients With Chronic Renal Failure Requiring Hemodialysis and Receiving Epoetin Maintenance Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EPOE-10-08
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2015-06

CONDITIONS: Chronic Renal Failure
Keywords: chronic renal failure requiring hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Epoetin Hospira administered IV for three doses (Experimental)
  Interventions: Drug: Epoetin Hospira
- Arm B: Epogen administered IV for three doses (Active Comparator)
  Interventions: Drug: Epogen

INTERVENTIONS:
Drug: Epoetin Hospira — IV dose 3 times a week.
  Arms: Arm A: Epoetin Hospira administered IV for three doses
Drug: Epogen — IV dose 3 times a week
  Arms: Arm B: Epogen administered IV for three doses

SUMMARY:
This study assessed the comparability of the pharmacokinetics (PK) of epoetin following intravenous administration of Hospira Epoetin and Epogen/Epoetin Alfa (Amgen) in patients with chronic renal failure receiving hemodialysis treatment.

DETAILED DESCRIPTION:
This is a multicenter, active-controlled, cross-over, evaluator-blind, Phase I study in patients with chronic renal failure requiring hemodialysis. The study comprises a 4-week Screening Period, a 1-week Pre-Treatment Period, a 1-week Treatment Period 1, a 1-week Treatment Period 2 and a Follow-up visit at Week 7.

Subject eligibility will be determined during the 4-week Screening Period. All subjects must be optimally titrated and stable to qualify for entry into Pre-Treatment Period.

During the 1-week Pre-treatment period the patients will continue on the same stable dose as they received during the Screening Period. Blood samples will be collected during the Pre-Treatment Period to assess pharmacokinetics of Epogen. Eligible subjects will be randomized at Day 1 of Treatment Period 1 to receive either Epoetin Hospira or Epogen (Amgen) by intravenous (IV) bolus injections administered three times a week for 1 week.

Subjects will then be switched to receive the alternate study drug for three times a week for 1 week in Treatment Period 2. Blood samples will be collected during Treatment periods 1 and 2 to assess pharmacokinetics of Epoetin Hospira and Epogen.

Primary endpoint, i.e. pharmacokinetics concentrations, will be evaluator blinded. After completing Treatment Period 2, all subjects will receive standard of care treatment and will undergo a Follow-up Visit at Week 7 (i.e., 28 days after Treatment Period 2).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent after risks and benefits of the study have been explained prior to any study related activities.
* Males and females between 18 and 75 years of age (both inclusive).
* Hemodialysis patients with chronic renal failure and anemia currently on stable epoetin treatment for at least 4 weeks prior to the Day 1 of Pre-treatment where during this period:

  * Epogen/Epoetin Alfa (Amgen) dose has been administered IV, 3 times a week and where each dose is <= 200 International Units(IU)/KG.
  * Hb levels were maintained within the 10-12 g/dL, with no more than a 0.5 g/dL change from the mean over this period.
  * No dose change during the last 4 weeks prior to Day 1 of pre-treatment period.
* Subjects on stable, adequate dialysis for at least 12 weeks prior to randomization, defined as no clinically relevant changes of dialysis regimen and/or dialyzer.
* Subjects with adequate iron stores, defined as serum ferritin >= 100 µg/L and transferrin saturation (TSAT) >20% prior to randomization.
* If female, subject must be postmenopausal for at lest 1 year prior to randomization, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or practicing at least one of the following forms of birth control:

  * hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to randomization.
  * intrauterine device (IUD)
  * double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream).

If hormonal contraceptives are used, the specific contraceptive must have been used for at least 3 months prior to randomization. If the subject is currently using a hormonal contraceptive, she should also use a barrier method during this study and for 1 month after last dose of Study Medication (Dosing Day 3 of Treatment Period 2).

Exclusion Criteria:

* A subject with any active, uncontrolled systemic disease that in the investigator's opinion may be significant to exclude participation in the study , including but not limited to microbial, viral or fungal infection or mental disease (including demyelinating diseases such as multiple sclerosis).
* History of drug abuse or alcohol abuse within 2 years prior to randomization as determined by the Investigator or a positive serum or saliva drug screen during the Screening Period or on Day 1 of each Treatment Period.
* Significant drug sensitivity or a significant allergic reaction to any drug, as well as known hypersensitivity or idiosyncratic reaction to epoetin (or it's excipients, including albumin) or any other related drugs.
* A subject who in the Investigator's opinion, has any clinically significant abnormal laboratory evaluations, including Human Immunodeficiency Virus (HIV), Hepatitis B virus surface antigen (HBsAg) and liver function taken at Screening Visit.
* Current treatment with long-acting epoetin analogues such as Aranesp.
* The following within 6 months prior to randomization: unstable congestive heart failure (New York Heart Association [NYHA] class III or IV), cerebrovascular accident, myocardial infarction, coronary angioplasty or by-pass surgery.
* Uncontrolled hypertension in Investigator's opinion within 4 weeks prior to randomization.
* A subject who has received a recent (within last 6 months) live or attenuated vaccination (except flu vaccination).
* A female subject who is pregnant, nursing, or planning a pregnancy during the study.
* Donated or lost >= 457 ml (i.e., 1 pint) blood volume (including plasmapheresis) or had a transfusion of any blood product within 3 months prior to randomization.
* Known clinically manifested untreated deficiency of folic acid and/or vitamin B12.
* Current participation or participation in a drug or other investigational research study within 30 days prior to randomization.
* May not be able to comply with the requirements of this clinical trial, communicate effectively with study personnel, or is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
* Known positive test for anti-epoetin antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted area under the serum epoetin concentration curve from the time of dose administration to 48 hours (AUC0-48) | On Day 1 and 2 of Pre-Treatment and Treatment Periods 1 and 2 predose (0 hour). On Day 3 of Pre-Treatment Period and Treatment Periods 1 and 2 (i.e., 3rd epoetin dose of the week) at predose (0 hour) and postdose (0.5, 1, 2, 4, 6, 8, 12, 24 and 48 hours)
Maximum serum epoetin concentration (Cmax) | On Day 1 and 2 of Pre-Treatment and Treatment Periods 1 and 2 predose (0 hour). On Day 3 of Pre-Treatment Period and Treatment Periods 1 and 2 (i.e., 3rd epoetin dose of the week) at predose (0 hour) and postdose (0.5, 1, 2, 4, 6, 8, 12, 24 and 48 hours)
AUC from time of dose administration to the time of the last measurable concentration (AUC0-t) | On Day 1 and 2 of Pre-Treatment and Treatment Periods 1 and 2 predose (0 hour). On Day 3 of Pre-Treatment Period and Treatment Periods 1 and 2 (i.e., 3rd epoetin dose of the week) at predose (0 hour) and postdose (0.5, 1, 2, 4, 6, 8, 12, 24 and 48 hours)
  If AUC0-48 cannot be calculated then AUC from time of dose administration to the time of the last measurable concentration (AUC0-t) will be used as the primary measure.

SECONDARY OUTCOMES:
Dose-adjusted Cmax | On Day 1 and 2 of Pre-Treatment and Treatment Periods 1 and 2 predose (0 hour). On Day 3 of Pre-Treatment Period and Treatment Periods 1 and 2 (i.e., 3rd epoetin dose of the week) at predose (0 hour) and postdose (0.5, 1, 2, 4, 6, 8, 12, 24 and 48 hours)
AUC from time of dose administration to the time of the last measurable concentration (AUC0-t) | On Day 1 and 2 of Pre-Treatment and Treatment Periods 1 and 2 predose (0 hour). On Day 3 of Pre-Treatment Period and Treatment Periods 1 and 2 (i.e., 3rd epoetin dose of the week) at predose (0 hour) and postdose (0.5, 1, 2, 4, 6, 8, 12, 24 and 48 hours)
Elimination rate Constant (λz) | On Day 1 and 2 of Pre-Treatment and Treatment Periods 1 and 2 predose (0 hour). On Day 3 of Pre-Treatment Period and Treatment Periods 1 and 2 (i.e., 3rd epoetin dose of the week) at predose (0 hour) and postdose (0.5, 1, 2, 4, 6, 8, 12, 24 and 48 hours)
Elimination halflife (t1/2) | On Day 1 and 2 of Pre-Treatment and Treatment Periods 1 and 2 predose (0 hour). On Day 3 of Pre-Treatment Period and Treatment Periods 1 and 2 (i.e., 3rd epoetin dose of the week) at predose (0 hour) and postdose (0.5, 1, 2, 4, 6, 8, 12, 24 and 48 hours)
Clearance (CL) | On Day 1 and 2 of Pre-Treatment and Treatment Periods 1 and 2 predose (0 hour). On Day 3 of Pre-Treatment Period and Treatment Periods 1 and 2 (i.e., 3rd epoetin dose of the week) at predose (0 hour) and postdose (0.5, 1, 2, 4, 6, 8, 12, 24 and 48 hours)
Volume of Distribution (Vd) | On Day 1 and 2 of Pre-Treatment and Treatment Periods 1 and 2 predose (0 hour). On Day 3 of Pre-Treatment Period and Treatment Periods 1 and 2 (i.e., 3rd epoetin dose of the week) at predose (0 hour) and postdose (0.5, 1, 2, 4, 6, 8, 12, 24 and 48 hours)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Downey, California
  - Tarzana, California
  - Denver, Colorado
  - Middlebury, Connecticut
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Gurnee, Illinois
  - Wichita, Kansas
  - Detroit, Michigan
  - Pontiac, Michigan
  - Minneapolis, Minnesota
  - Gulfport, Mississippi
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Knoxville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Alexandria, Virginia